CLINICAL TRIAL: NCT04630730
Title: Intravesical Recombinant BCG (Bacillus Calmette Guérin) Followed by Perioperative Chemo-immunotherapy for Patients With Muscle-invasive Bladder Cancer (MIBC). A Multicenter, Single-arm Phase II Trial
Brief Title: Intravesical Recombinant BCG Followed by Perioperative Chemo-immunotherapy for Patients With MIBC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 06/19
Record Dates: First submitted 2020-11-06; First posted 2020-11-16 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Bladder Cancer
Keywords: muscle-invasive bladder cancer; MIBC; intravesical BCG; Bacillus Calmette Guérin; VPM1002BC; atezolizumab; Cisplatin; Gemcitabine; neoadjuvant; adjuvant
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — atezolizumab; Cisplatin; Gemcitabine

STUDY DESIGN:
Intervention Model Description: Prospective single-arm open-label multicenter phase II trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recombinant intravesical BCG (Experimental): The Intravesical recombinant BCG (Bacillus Calmette-Guérin - VPM1002BC) is used as an immuno-stimulating agent. The patient will receive 3 weekly BCG instillations as induction treatment.
  4 cycles of atezolizumab, a fully humanized, engineered monoclonal antibody of IgG1 isotype against the protein programmed cell death-ligand 1 (PD-L1 inhibitor) will be administered in combination with the standard neoadjuvant chemotherapy cisplatin/gemcitabine.
  After surgery atezolizumab will be administered in the adjuvant setting for 13 cycles.
  Interventions: Drug: Recombinant intravesical BCG (Bacillus Calmette-Guérin VPM1002BC); Drug: Atezolizumab; Drug: Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Recombinant intravesical BCG (Bacillus Calmette-Guérin VPM1002BC) — 1 dose of VPM1002BC, live, 1-19.2 x 108 colony forming units (CFU) on day 1, 8 (+/- 1 day) and 15 (+/- 1 day)
  Other Names: VPM1002BC
Drug: Atezolizumab — Neoadjuvant immunotherapy with atezolizumab, 4 cycles 1200 mg fixed dose iv infusion on d1 q3w starting 4-16 weeks after date of surgery
  Other Names: Tecentriq™
Drug: Cisplatin — Neoadjuvant chemotherapy with cisplatin: 4 cycles 70mg/m2 iv infusion on d1 q3w (starting on d22)
  Other Names: Platinol®
Drug: Gemcitabine — Neoadjuvant chemotherapy with gemcitabine: 4 cycles 1000 mg/m2 iv infusion on d1 and d8 q3w (starting on d22)
  Other Names: Gemzar ®

SUMMARY:
Current treatment of localized muscle-invasive bladder cancer is still associated with high relapse and death rate as well as the need for complete bladder resection or irradiation.

The primary objective of this trial is to increase the rate of pathologic complete remission (pCR) at the time of radical cystectomy by the combination of local bladder instillation with Bacillus Calmette Guérin (BCG) in combination with systemic immunotherapy with atezolizumab and standard chemotherapy with cisplatin/gemcitabine.

The trial tests the hypothesis whether BCG can enhance systemic and local immune response and thereby increase pCR rate and consequently also event-free survival. Improving pCR rate would be a next step to the ultimate goal of omitting radical surgery or extensive local radiotherapy to the bladder for these patients.

DETAILED DESCRIPTION:
Current treatment of localized muscle-invasive bladder cancer is still associated with high relapse and death rate as well as the need for complete bladder resection or irradiation.

In recent years, immunotherapy using PD-1 or PD-L1 immune checkpoint inhibitors (ICI) proved successful for patients with metastatic bladder cancer. The checkpoint inhibitors atezolizumab (anti PD-L1), pembrolizumab (anti PD-1) and nivolumab (anti PD-1) now represent the standard of care in the second line setting of metastatic bladder cancer and are all approved by Swissmedic for this indication.

First results, in 2018, have been presented and published using immune checkpoint inhibitors as neoadjuvant treatment for localized muscle-invasive bladder cancer. SAKK has also performed a single arm phase II trial using neoadjuvant chemo-immunotherapy with cisplatin/gemcitabine in combination with the PD-L1 inhibitor durvalumab (SAKK 06/17). A preplanned interim analysis of the first 30 operated patients revealed a pCR rate of 30%. In this study, residual non-muscle invasive bladder cancer (NMIBC) was found in approximately 15% of cases. While these results are encouraging, the improvement of pCR rate compared to cisplatin-based chemotherapy alone is small and further improvement is needed.

BCG induces an intense local inflammatory response that mediates tumor immunity. Several steps are involved in mounting the inflammatory response including attachment to the urothelium with uptake by antigen presenting cells (APC) and putative internalization into urothelial cells followed by a boost of the innate immune response and induction of adaptive responses. Based on these findings, intravesical BCG appears to be a very interesting agent to enhance the immune response and act as an adjuvant agent to increase anti-tumor response with immune checkpoint inhibition using monoclonal antibodies such as atezolizumab. The combination of intravesical BCG and systemic immune checkpoint inhibition is being studied for patients with non-muscle invasive bladder cancer in several ongoing phase III trials.

the investigators therefore propose to add an induction cycle of intravesical recombinant BCG (VPM1002BC) (total of 3 weeks) to the backbone of neoadjuvant chemo-immunotherapy with cisplatin/gemcitabine and atezolizumab. The trial tests the hypothesis if recombinant BCG can enhance systemic and local immune response and thereby increase pCR rate and consequently also event-free survival. Improving pCR rate would be a next step to the ultimate goal of omitting radical surgery or extensive local radiotherapy to the bladder for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to ICH/GCP regulations before registration and prior to any trial specific procedures
* Histologically proven urothelial cell carcinoma of the bladder (cT2, cT3 or cT4a and ≤ cN1 (defined as a solitary lymph node ≤ 2 cm in the greatest dimension) and cM0) and be considered suitable for curative multimodality treatment including radical cystectomy by a multidisciplinary tumor board
* All histological subtypes eligible with the exception of small cell component
* Age ≥ 18 years
* WHO performance status 0-1
* Hematological function: hemoglobin ≥ 90 g/L, neutrophils ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L
* Hepatic function: total bilirubin ≤ 1.5 x ULN (except for patients with Gilbert's disease ≤ 3.0 x ULN), AST ≤ 2.5 x ULN and ALT ≤ 2.5 x ULN, AP ≤ 2.5 x ULN
* Renal function: estimated glomerular filtration rate (eGFR) > 50 mL/min/1.73m², according to CKD-EPI formula
* Women of childbearing potential must use effective contraception, are not pregnant or lactating and agree not to become pregnant during trial treatment and until 5 months after the last dose of investigational drug
* Men agree not to donate sperm or to father a child during trial treatment and until 5 months after the last dose of investigational drug (www.swissmedicinfo.ch).

Exclusion Criteria:

* Any pathological evidence of small-cell carcinoma component
* Presence of any distant metastasis
* History of hematologic or primary solid tumor malignancy, unless in remission for at least 3 years after registration, with the exception of adequately treated cervical carcinoma in situ, localized non-melanoma skin cancer or low risk localized prostate cancer (T1-T2a, Gleason <7, PSA <10ng/ml)
* Residual urinary bladder volume after micturition > 150ml (measured by ultrasound of bladder or inserted catheter)
* Prior treatment for bladder cancer including BCG instillations. Single dose intravesical chemotherapy instillation after TURB is allowed
* Bladder surgery or traumatic catheterization or TURB within 14 days prior to the expected start of BCG trial treatment
* Uncontrollable urinary tract infection, macroscopic haematuria, suspicion of bladder perforation, urethral strictures (if interfering with trial procedures)
* Any conditions preventing the patient from keeping BCG instillation in the bladder for at least 1 hour; anticholinergics are allowed to achieve this criterion
* Any previous treatment with a PD-1 or PD-L1 inhibitor, including atezolizumab
* Concomitant or prior use of immunosuppressive medication within 28 days before registration, with the exceptions of intranasal and inhaled corticosteroids, or systemic corticosteroids which must not exceed 10 mg/day of prednisone (or a dose equivalent corticosteroid) and the premedication for chemotherapy
* Concurrent treatment with other experimental drugs or other anticancer therapy, treatment in a clinical trial within 28 days prior to registration
* Major surgical procedure within 28 days prior to registration
* Preexisting peripheral neuropathy (> grade 1)
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

  * Patients with vitiligo or alopecia
  * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Patients without active disease in the last 5 years may be included but only after consultation with the Coordinating Investigator
  * Patients with celiac disease controlled by diet alone
* Known history of human immunodeficiency virus (HIV) or active chronic Hepatitis C or Hepatitis B Virus infection or any uncontrolled active systemic infection requiring intravenous (iv) antimicrobial treatment
* Known history of tuberculosis, known history of primary immunodeficiency, known history of allogeneic organ transplant, or receipt of live attenuated vaccine within 4 weeks prior to registration, or anticipation of need for such a vaccine during atezolizumab treatment or within 5 months after the final dose of atezolizumab
* Severe or uncontrolled cardiovascular disease (congestive heart failure NYHA III or IV), unstable angina pectoris, history of myocardial infarction within the last six months, serious arrhythmias requiring medication (with exception of atrial fibrillation or paroxysmal supraventricular tachycardia), significant QT-prolongation, uncontrolled hypertension
* Any concomitant drugs contraindicated for use with the trial drugs according to the approved product information
* Known hypersensitivity to trial drugs or to any component of the trial drugs
* Any other serious underlying medical, psychiatric, psychological, familial or geographical condition, which in the judgment of the investigator may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment-related complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2022-06-24 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Pathological complete remission (pCR) | At the date of tumor assessment after surgery, estimated at approximately 20 to 24 weeks after treatment start
  The primary endpoint of the trial is pCR after neoadjuvant treatment defined as ypT0ypN0 and no evidence of non-muscle invasive bladder cancer (low grade, high grade or CIS).
  The primary analysis will be based on the results from central pathology review.

SECONDARY OUTCOMES:
Event-free survival (EFS) | From the date of treatment start until the date of progressive disease, recurrence of locoregional disease, appearance of metastases or death, whichever occurs first, assessed up to 5 years after surgery
  EFS is defined as the time from treatment start until one of the following events, whichever comes first:
  * Progression during neoadjuvant treatment leading to inoperability
  * Recurrence or progression (in case of disease persistence) of locoregional disease after surgery
  * Appearance of metastases at any localization
  * Death Patients without event at the time of analysis and patients starting a subsequent treatment in the absence of an event will be censored at the date of the last available assessment showing no event before the start of the subsequent treatment, if any.
  This endpoint will be calculated for patients in the FAS.
Recurrence-free survival (RFS) after R0 resection | From the date of surgery until the date recurrence of locoregional disease, appearance of metastases or death, whichever occurs first, assessed up to 5 years after surgery
  RFS after R0 resection is defined as the time from surgery until one of the following events, whichever comes first:
  * Recurrence of locoregional disease
  * Appearance of metastases at any localization
  * Death Patients without event at the time of analysis and patients starting a subsequent treatment in the absence of an event will be censored at the date of the last available assessment showing no event before the start of the subsequent treatment, if any.
  This endpoint will only be calculated for patients in the R0 resection set.
Overall survival (OS) | From the date of treatment start until the date of death, assessed up to 5 years after surgery
  OS is defined as the time from treatment start until death from any cause. Patients not experiencing an event will be censored at the last date they were known to be alive.
  This endpoint will be calculated for patients in the FAS.
Quality of resection: Complete resection | At the date of tumor assessment after surgery, estimated at approximately 20 to 24 weeks after treatment start
  The quality of resection will be assessed in the following way:
  • Complete resection (R0) defined as free resection margins proved microscopically This endpoint will only be calculated for patients in the resected patients set.
Quality of resection: Completeness of the lymphadenectomy and surgery | At the date of tumor assessment after surgery, estimated at approximately 20 to 24 weeks after treatment start
  The quality of resection will be assessed in the following way:
  • Completeness of the lymphadenectomy and surgery using the photo documentation and histopathology This endpoint will only be calculated for patients in the resected patients set.
Quality of resection: Postoperative complications | At the date of tumor assessment after surgery, estimated at approximately 20 to 24 weeks after treatment start
  The quality of resection will be assessed in the following way:
  • Postoperative complications will be assessed using the Clavien-Dindo classification.
  This endpoint will only be calculated for patients in the resected patients set.
Pathological response (PaR) rate | At the date of tumor assessment after surgery, estimated at approximately 20 to 24 weeks after treatment start
  PaR rate is defined as pathological downstaging to ≤ ypT1N0M0. The proportion of patients with PaR will be calculated for patients in the resected patients set.
  This endpoint will only be calculated for patients in the resected patients set.
Pattern of recurrence | at the date of the first occurrence of recurrence, assessed up to 5 years after surgery
  Pattern of recurrence is defined as location of first tumor recurrence. Patterns can be locoregional or distant or any combination of these patterns.
  Patients with secondary malignancies or patients with no recurrence will not be taken into consideration for this endpoint.
Treatment feasibility | from the date of treatment start until the date of treatment stop, estimated at approximately 63 to 79 weeks after treatment start
  The following feasibility criteria will be assessed:
  * Completion of 3 instillations of intravesical VPM1002BC
  * Completion of 4 cycles of neoadjuvant chemotherapy
  * Completion of 4 cycles of neoadjuvant atezolizumab treatment
  * Timely admission to and completion of planned surgery
  * Timely initiation and completion of 13 cycles of adjuvant atezolizumab treatment
Adverse events | from the date of registration until 28 days after the date of treatment stop, estimated at approximately 67 to 83 weeks after treatment start
  All AEs will be assessed according to NCI CTCAE v5.0. This endpoint will be calculated for patients in the safety set.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Cathomas, MD, Study Chair — Kantonsspital Graubünden, Chur
Locations (10):
- Switzerland (10):
  - Klinik Hirslanden - Onkozentrum Hirslanden, Zurich, Canton of Zurich
  - Kantonsspital Baden, Baden
  - Universitaetsspital Basel, Basel
  - Istituto Oncologico della Svizzera Italiana - Ospedale Regionale Bellinzona e Valli, Bellinzona
  - Lindenhofspital, Bern
  - Kantonsspital Graubuenden, Chur
  - Hôpitaux Universitaires Genève HUG, Geneva
  - Luzerner Kantonsspital, Lucerne
  - Kantonsspital St. Gallen, Sankt Gallen
  - UniversitaetsSpital Zuerich, Zurich

REFERENCES:
- [Derived] Petrausch U, Spahn M, Schneider M, Hayoz S, Rentsch CA, Rothschild S, Omlin A, Cathomas R. Novel sequential treatment strategy for patients with muscle-invasive bladder cancer (MIBC): intravesical recombinant BCG, followed by neoadjuvant chemoimmunotherapy, radical cystectomy plus pelvic lymphadenectomy and adjuvant immunotherapy - protocol of a multicentre, single arm phase 2 trial (SAKK 06/19). BMJ Open. 2023 Jun 7;13(6):e067634. doi: 10.1136/bmjopen-2022-067634. PMID 37286312